CLINICAL TRIAL: NCT02265159
Title: Intervention Trial Evaluating Focal Therapy Using High Intensity Focused Ultrasound for the Treatment of Prostate Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Daniel Eberli, PD Dr. med. PhD, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2013-0415
Record Dates: First submitted 2014-09-29; First posted 2014-10-15 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal Therapy Using High Intensity Focused Ultrasound (Other)
  Interventions: Procedure: Focal Therapy Using High Intensity Focused Ultrasound

INTERVENTIONS:
Procedure: Focal Therapy Using High Intensity Focused Ultrasound
  Other Names: Focal HIFU

SUMMARY:
The investigators aim to evaluate cancer control, genitourinary, rectal and overall health-related quality of life outcomes and effectiveness of focal therapy for localised prostate cancer using High Intensity Focused Ultrasound (HIFU).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer on trans-rectal or transperineal template prostate biopsies
* Template biopsy:

  * unilateral disease (Gleason ≤4+3)
  * bilateral disease: presence of clinically significant cancer in both sides (Gleason ≤4+3) OR clinically insignificant disease with a burden of >50% of biopsy cores taken on that side, OR bilateral clinically insignificant disease and <50% of biopsy cores positive on any one side but with dominant disease burden on one side
* Stage T1-T2cN0M0 disease, as determined by local guidelines (radiological T3a permitted)
* Serum PSA ≤15
* Life expectancy of ≥10 years
* Signed informed consent by patient
* An understanding of the German language sufficient to understand written and verbal information about the trial and consent process

Exclusion Criteria:

* Men who have had androgen suppression/hormone treatment within the previous 12 months for their prostate cancer
* Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging
* Men with an inability to tolerate a transrectal ultrasound
* Men with latex allergies as the HIFU probe is covered with a latex condom sheath prior to insertion into the back passage
* Men who have undergone prior significant rectal surgery preventing insertion of trans-rectal HIFU probe (decided on the type of surgery in individual cases)
* Men who have had previous HIFU, cryosurgery, thermal or microwave therapy to the prostate.
* Men who have undergone a Transurethral Resection of the Prostate (TURP) for symptomatic lower urinary tract symptoms within 6 months. These patients may be included within the trial if deferred from consenting and screening until at least 6 months following the TURP.
* Men not fit for major surgery as assessed by a Consultant Anaesthetist
* Men unable to have pelvic MRI scanning (severe claustrophobia, permanent cardiac pacemaker, metallic implant etc likely to contribute significant artefact to images)
* Presence of metal implants/stents in the urethra
* Presence of prostatic calcification and cysts (on transrectal ultrasound) whose location will interfere with effective delivery of HIFU therapy
* Men with renal impairment with a glomerular filtration rate of <35ml/min (unable to tolerate Gadolinium dynamic contrast enhanced MRI).

Ages: 40 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Oncological safety | 36 months
  To determine the proportion of men who are free of clinically significant prostate cancer in the treated area AND are free of clinically significant prostate cancer in the untreated area 36 months after focal therapy using HIFU
Oncological safety | 36 months
  To determine the proportion of men who are free of any prostate cancer in the treated area AND are free of clinically significant prostate cancer in the untreated area 36 months after focal therapy using HIFU

SECONDARY OUTCOMES:
Biochemical failure | 36 months
  To analyse the rate of biochemical recurrence by measuring PSA values following focal therapy using HIFU:
  * biochemical recurrence defined according to the Phoenix Consensus OR
  * by PSA velocity >1 ng/ml/year OR PSA doubling time </=3 years
Sensitivity and specificity of MRI imaging | 36 months
  To determine the clinical validity (area under the receiver operating characteristics curve (AUC), sensitivity, specificity, negative and positive predictive values, inter-observer variability) of
  * multi-parametric MR-imaging to predict presence of clinically significant prostate cancer on transperineal template prostate mapping biopsies prior to focal therapy
  * MR-imaging changes to predict presence of residual/recurrent clinically significant prostate cancer on biopsy
Health care costs | 36 months
  To determine the costs of treatment and longitudinal morbidity associated with complications at 36 months compared to other treatments of localized prostate cancer.
Erectile function | 36 months
  Rate of erectile dysfunction and time to return of erectile function (measured by the IIEF-15)
Orgasmic function | 36 months
  Rate of loss of ejaculation and orgasm (measured by the IIEF-15)
Sexual function | 36 months
  Rate of pain during intercourse
Erectile function | 36 months
  Number of men using phosphodiesterase-5 inhibitors to maintain erectile function (measured by the IIEF-15)
Continence | 36 months
  Rate of urinary incontinence (pad free, leak free and padfree alone) (determined by the UCLA-EPIC urinary continence questionnaire)
Continence | 36 months
  Time to return of continence (pad free, leak free and padfree alone) (determined by the UCLA-EPIC urinary continence questionnaire)
Lower urinary tract symptoms | 36 months
  Rate of lower urinary tract symptoms (as determined by IPSS scores)
Bowel function | 36 months
  Rate of bowel toxicity (determined by the UCLA-EPIC Bowel questionnaire )
Anxiety | 36 months
  Anxiety levels (measured by the Hospital Anxiety and Depression Scale and Memorial Anxiety Scale for Prostate Cancer
Quality of life | 36 months
  General health related quality of life (measured using FACT-P Version 4 )
General histological outcome | 36 months
  To determine the histological outcomes at 6, 12 and 36 months
Secondary intervention | 36 months
  Rate of secondary prostate cancer intervention (prostatectomy, radiotherapy, androgen ablation)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eberli, PD Dr. PhD, Principal Investigator — Klinik für Urologie, Universitätsspital Zürich
Locations (1):
- Klinik für Urologie, Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland